CLINICAL TRIAL: NCT04863846
Title: Development and Implementation of an Evidence-based Clinical Algorithm for the Expected Difficult Intubation
Brief Title: Evidence-based Algorithm for the Expected Difficult Intubation
Acronym: Expect-it
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-10459-BO-ff
Record Dates: First submitted 2021-04-13; First posted 2021-04-28 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Airway Management; Intubation, Intratracheal
Keywords: Laryngoscopy; Laryngoscopes; Diagnostic Techniques, Respiratory System
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinical standard (first study phase): Current clinical standard, non-algorithm-based decision-making (prior to implementation of the algorithm)
  Interventions: Other: No intervention, observational study
- Algorithm-based allocation (second study phase): New algorithm-based allocation to an intubation technique (after implementation of the algorithm)
  Interventions: Other: No intervention, observational study

INTERVENTIONS:
Other: No intervention, observational study — Exposure of interest: clinical implementation of an algorithm

SUMMARY:
The Expect-it study aims to accompany the development and clinical implementation process of a new algorithm for the management of expected difficult intubation. The new algorithm is designed to allocate patients to specific tracheal intubation techniques. After assessing the status quo (non-algorithm-based decision-making) the new algorithm-based allocation will be compared with this clinical standard within a confirmatory diagnostic accuracy study (post-implementation).

DETAILED DESCRIPTION:
Difficult tracheal intubation is one of the major reasons for anesthesia-related adverse events. Patients undergoing ear, nose & throat (ENT) or oral and maxillofacial (OMS) surgery often require tracheal intubation for general anesthesia but are at increased risk for difficult tracheal intubation. Currently, existing preoperative tests for the prediction of difficult intubation show low diagnostic accuracy. Moreover, as the results of these prediction tests are not coupled with concrete treatment recommendations, they cannot be used targeted within preventive concepts. An evidence based rational algorithm for the management of expected difficult intubation has not been developed yet. It is unknown, if an algorithm-based allocation to an intubation approach might be advantageous compared with a non-algorithm-based allocation strategy.

The Expect-it study aims to accompany the development and clinical implementation process of a new algorithm for the management of expected difficult intubation. This new algorithm is designed to provide an evidence-based decision-making tool for a rational pre-choice of tracheal intubation techniques, anesthetized intubation by direct laryngoscopy (DL) or videolaryngoscopy (VL) or awake tracheal intubation (ATI). In the first study phase the status quo (clinical standard, non-algorithm-based decision-making) will be assessed (three-month period with an approximated case number of up to 600 patients). The Expect-it algorithm will be implemented thereafter. Between both study phases, the algorithm will be updated (based on the findings of the first phase), sensitivity and specificity of the clinical standard will be calculated, sample size will critically be appraised and readjusted (approximately 600 within at least three months), if appropriate. The second study phase is a confirmatory diagnostic accuracy study for the new algorithm with a single test study design, that aims to proof, if the new Expect-it algorithm is superior or at least non-inferior to the clinical standard, defined as superiority in either the specificity or sensitivity and non-inferiority in the other co-primary endpoint in each domain (ATI, DL, VL) (pre-planned preliminary analysis of the first study phase; IRB amendment 2021-10459_2-BO-ff, December 3, 2021). Sensitivity and specificity are considered co-primary endpoints. Study planning and conduction is in accordance with the Standards for Reporting Diagnostic accuracy studies (STARD) statement. The Expect-it study will further include two surveys among anesthetist in the study center in order to evaluate challenges and obstacles associated with the implementation process and possible clinical implications of the algorithm. An additional analysis will be performed to test a core data set for an 'anesthesia alert card'.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ENT or OMS surgery that require general anesthesia with tracheal intubation (either DL, VL or ATI)
* Age ≥ 18 years

Exclusion Criteria:

* Denial of consent
* Planned intubation technique is not designated in the study protocol as it differs from either DL, VL, ATI (e.g. primary tracheotomy or rigid bronchoscopy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive sampling: Adult patients that undergo ENT or OMS surgery in a tertiary care hospital who require tracheal intubation and consent to participate within two predefined study periods of at least 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 1282 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-01-29 (Actual); Study Completion 2022-01-29 (Actual)

PRIMARY OUTCOMES:
First phase: sensitivity and specificity (co-primary endpoints) of the clinical standard | 3 months
  Clinical assessment
Second phase: sensitivity and specificity (co-primary endpoints) of 'ATI recommendation' by the algorithm vs. 'VL/DL' | 3 months
  Clinical assessment
Second phase: sensitivity and specificity (co-primary endpoints) of 'DL recommendation' by the algorithm vs. 'VL/ATI' | 3 months
  Clinical assessment
Second phase: sensitivity and specificity (co-primary endpoints) of 'VL recommendation' by the algorithm vs. 'DL/ATI' | 3 months
  Clinical assessment

SECONDARY OUTCOMES:
Post-intubation recommendation for an intubation method | 1 hour
  Recommendation of the responsible anesthetist
Post-intubation recommendation for an anesthesia alert card | 1 hour
  Recommendation of the responsible anesthetist
Post-intubation diagnosis 'difficult intubation' | 1 hour
  Rating of the responsible anesthetist
Post-intubation diagnosis 'difficult face-mask-ventilation' | 1 hour
  Rating of the responsible anesthetist
Classification of intubation difficulty (VIDIAC classification) | 1 hour
  Rating between -1 and 5 points
Best glottic view | 1 hour
  Grading according to 'Percentage of Glottis Opening' (POGO)
Best glottic view | 1 hour
  Grading according to the Cormack Lehane classification (I-IV)
First pass success rate | 1 hour
  Percentage of successful intubations with one attempt
Overall success rate of the first choice technique | 1 hour
  Percentage of successful intubation without transition to another technique
Number of attempts | 1 hour
  Total number of attempts until airway established
Intubation time | 1 hour
  Time to successful tracheal intubation
Lowest oxygen saturation | 1 hour
  Measured with pulse oxymetry during anesthesia induction
Overall intubation difficulty, ease of intubation, quality of visualization | 1 hour
  Subjective ratings on visual analogue scales (0 to 100 with 0 being the best)
Airway-related adverse events | 1 hour
  Laryngospasm, bronchospasm, larynx trauma, airway trauma, soft tissue trauma, oral bleeding, edema, dental damage, corticosteroid application, accidental esophageal intubation, aspiration, hypotension or hypoxia
Patient discomfort, satisfaction, symptoms | 12 hours
  Clinical assessment during follow-up
Clinical evaluation of a core dataset 'anesthesia alert card' | 10 months
  Rating of various anesthetist
Quality of care of the current clinical standard and the effects of algorithm implementation | 7 months
  Survey among anesthetist

CONTACTS AND LOCATIONS:
Overall Officials: Martin Petzoldt, MD, Study Chair — Universitätsklinikum Hamburg-Eppendorf; Antonia Zapf, PhD, Study Chair — Universitätsklinikum Hamburg-Eppendorf; Christian Zöllner, MD, Study Chair — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany